CLINICAL TRIAL: NCT02750800
Title: Post-marketing Observational Study to Evaluate the Effect of HUMIRA (Adalimumab) Treatment With AbbVie's Patient Support Program on Patient Reported Outcomes and Health Resource Utilization in Inflammatory Arthritis, Psoriasis and Inflammatory Bowel Diseases in Hungary in a Real-life Setting: VALUE
Brief Title: Post-marketing Observational Study to Evaluate the Incremental Impact of AbbVie's Patient Support Program on Patient Reported Outcomes and Health Resource Utilization in Inflammatory Arthritis, Psoriasis and Inflammatory Bowel Diseases in Hungary (VALUE)
Acronym: VALUE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-673
Record Dates: First submitted 2016-04-13; First posted 2016-04-26 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Psoriasis; Crohn's Disease; Ulcerative Colitis
Keywords: Rheumatoid arthritis; Ankylosing spondylitis; Psoriatic arthritis; Psoriasis; Crohn's disease; Ulcerative colitis; Patient support program; Quality of life; Patient related outcomes; Observational study; Adalimumab; Humira; Adherence; Health-related quality of life; Healthcare resource utilization; Disease activity; Treatment satisfaction; Workability
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Psoriasis; Crohn Disease; Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adalimumab and AbbVie Care 2.0: Adalimumab administered via subcutaneous (SC) injection for 12 months according to the approved EMA label and Hungarian financial protocols and supportive services via the AbbVie Care 2.0 patient support program
  Interventions: Biological: Adalimumab; Behavioral: AbbVie Care 2.0

INTERVENTIONS:
Biological: Adalimumab — Pre-filled syringe or pen, administered by subcutaneous injection
  Other Names: Humira; ABT-D2E7
Behavioral: AbbVie Care 2.0 — Supportive services provided to participants included reminder calls, emails, text messages, nursing services, dietician, and psychological support. An adalimumab starter pack, injection guide, digital and print educational materials were also provided.

SUMMARY:
The objective of this post-marketing observational study (PMOS) was to evaluate the effectiveness of adalimumab plus the AbbVie Care 2.0 patient support program in participants with rheumatoid arthritis (RA), ankylosing spondylitis (AS), psoriatic arthritis (PsA), psoriasis (Ps), Crohn's disease (CD) or ulcerative colitis (UC) in the routine clinical setting in Hungary.

DETAILED DESCRIPTION:
This was a prospective, open label, multicenter, observational cohort study. Adalimumab was prescribed in the usual manner in accordance with the terms of the local marketing authorization and professional and reimbursement guidelines with regards to dose, population and indication. AbbVie offered an array of services as part of a patient support program, called AbbVie Care 2.0, to study participants. The purpose of the AbbVie Care 2.0 program was to provide educational resources that aimed to help participants understand their health condition and disease management (e.g., lifestyle - exercise or diet), but also help to them understand how to administer the product safely and be empowered to stay on track with their prescribed treatment plan, all with the goal of maximizing patient outcomes. There were five target visits: a baseline visit at enrollment and follow-up visits at 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of rheumatoid arthritis (RA), ankylosing spondylitis (AS), psoriatic arthritis (PsA), psoriasis (Ps), Crohn's disease (CD) or ulcerative colitis (UC) by the treating physician
* Age ≥ 18 years at the time of enrollment
* RA, AS, PsA, Ps, UC or CD patients for whom adalimumab treatment was indicated as per local Summary of Product Characteristics (SmPC) and professional/reimbursement guidelines
* Participants assigned to adalimumab treatment not more than 1 month prior to inclusion
* Participants to whom participation in AbbVie Care 2.0 Patient Support Program (PSP) program was offered and participant decided to join and had started the PSP
* Participants willing to be involved in the study and to sign patient informed consent form (ICF) and subject information form (SIF) in order to allow use and disclosure of his/her personal health information

Exclusion Criteria:

* Participants who could not be treated with adalimumab according to the local adalimumab SmPC and local professional and reimbursement guidelines
* Participants treated with > 1 prior biologic disease modifying anti rheumatic drug (DMARD) for RA, AS, PsA, Ps, UC or CD
* Prior treatment with adalimumab for more than 1 month
* Participants currently participating in other clinical research studies
* Participants who were unwilling or unable to complete the quality of life and other patient-reported questionnaires

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with rheumatoid arthritis (RA), ankylosing spondylitis (AS), psoriatic arthritis (PsA), psoriasis (Ps), Crohn's disease (CD) or ulcerative colitis (UC)
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Morisky DE, Malotte CK, Choi P, Davidson P, Rigler S, Sugland B, Langer M. A patient education program to improve adherence rates with antituberculosis drug regimens. Health Educ Q. 1990 Fall;17(3):253-67. doi: 10.1177/109019819001700303. PMID 2228629
- [Background] Morisky DE, DiMatteo MR. Improving the measurement of self-reported medication nonadherence: response to authors. J Clin Epidemiol. 2011 Mar;64(3):255-7; discussion 258-63. doi: 10.1016/j.jclinepi.2010.09.002. Epub 2010 Dec 8. No abstract available. PMID 21144706
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set: participants who met all of the inclusion criteria and none of the exclusion criteria and received at least one dose of adalimumab
Period: Overall Study
Arm/Group | Adalimumab and AbbVie Care 2.0
Started | 412
Completed | 314
Not Completed | 98
Not completed — Adverse Event | 18
Not completed — Lost to Follow-up | 12
Not completed — Investigator decision | 53
Not completed — Patient request | 12
Not completed — Other, not specified | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants who met all of the inclusion criteria and none of the exclusion criteria and received at least one dose of adalimumab
Groups:
- Ankylosing Spondylitis: Participants with ankylosing spondylitis
- Crohn's Disease: Participants with Crohn's disease
- Psoriasis: Participants with psoriasis
- Psoriatic Arthritis: Participants with psoriatic arthritis
- Rheumatoid Arthritis: Participants with rheumatoid arthritis
- Ulcerative Colitis: Participants with ulcerative colitis
- Total: Total of all reporting groups
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis | Total
Number analyzed (Participants) | 76 | 62 | 69 | 75 | 67 | 63 | 412
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing data for one participant with Crohn's disease and one participant with ulcerative colitis
  years
    number analyzed (Participants) | 76 | 61 | 69 | 75 | 67 | 62 | 410
    (all) | 47.8 (13.33) | 35.5 (12.10) | 51.7 (14.24) | 50.6 (11.29) | 52.7 (10.44) | 37.6 (12.52) | 46.4 (14.00)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data for one participant with ulcerative colitis
  Participants
    number analyzed (Participants) | 76 | 62 | 69 | 75 | 67 | 62 | 411
    Female | 29 | 31 | 22 | 34 | 53 | 27 | 196
    Male | 47 | 31 | 47 | 41 | 14 | 35 | 215
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Short Form 36 Version 2.0 (SF-36 V2) Physical Component Summary (PCS) Score at 12 Months
Description: The health assessment questionnaire Short Form 36 Version 2.0 (SF-36 V2 ) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5-8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 "worst"-100 "best"). Positive numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 60 | 49 | 51 | 55 | 48 | 44
units on a scale | 11.02 (10.24) | 7.63 (9.51) | 4.38 (9.14) | 12.26 (10.73) | 11.81 (10.83) | 9.02 (8.65)

2. Secondary Outcome: Mean Change From Baseline in Short Form 36 Version 2.0 (SF-36 V2) Mental Component Summary (MCS) Score at 12 Months
Description: as for outcome 1
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 60 | 49 | 51 | 55 | 48 | 44
units on a scale | 9.63 (13.31) | 10.60 (15.87) | 6.61 (13.25) | 8.54 (12.63) | 5.99 (11.86) | 11.50 (15.35)

3. Secondary Outcome: Mean Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Index Score at 12 Months
Description: The EQ-5D-5L measures quality of life in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on five levels of severity (1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, 5: extreme problems), and a separate visual analog scale (VAS). Responses to the five dimension scores were combined and converted into a single preference-weighted health utility index score. The range for the EQ-5D-5L index score is 0 to 1 with '0' defined as a health state equivalent to being dead and '1' is full health. The higher the score the better the health status. Positive numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 59 | 48 | 55 | 56 | 54 | 46
units on a scale | 0.185 (0.18) | 0.169 (0.19) | 0.084 (0.14) | 0.203 (0.18) | 0.152 (0.19) | 0.123 (0.14)

4. Secondary Outcome: Mean Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale Score at 12 Months
Description: The EQ-5D-5L measures quality of life in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on five levels of severity (1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, 5: extreme problems), and a separate visual analog scale (VAS). Participants rated their health on a vertical visual analogue scale, where the endpoints were labelled 100, "The best health you can imagine"and 0, "The worst health you can imagine". Positive numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 59 | 48 | 55 | 56 | 55 | 44
units on a scale | 18.5 (29.23) | 22.2 (22.65) | 11.4 (20.50) | 29.7 (28.52) | 22.6 (33.82) | 25.1 (26.11)

5. Secondary Outcome: Mean Change From Baseline in Short Quality of Life in Inflammatory Bowel Disease Questionnaire (SIBDQ) Score at 12 Months in Participants With Crohn's Disease and Ulcerative Colitis
Description: The SIBDQ is a disease-specific health-related quality of life (HRQOL) questionnaire, able to detect and define meaningful clinical changes in inflammatory bowel disease (IBD) participants by measuring physical, social and emotional status. The SIBDQ consists of 10 questions; each question is scored on a scale from 1 (poor QOL) to 7 (optimum QOL). A higher score indicates a better health-related quality of life. Total scores range from 10 (poor QoL) to 70 (good QoL). Positive numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with either Crohn's disease or ulcerative colitis and evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 49 | 46
units on a scale | 11.6 (17.5) | 16.1 (16.6)

6. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI) Score at 12 Months in Participants With Psoriasis and Psoriatic Arthritis
Description: The Dermatology Life Quality Index (DLQI) is a self-reported questionnaire for capturing psychosocial effects of chronic skin disease on different areas of life within the previous seven days. The ten questions cover six areas: symptoms/feelings, daily activities, leisure, work/school, personal relationship, effects of treatment on daily life. Total DLQI scores range from 0 to 30, with 0 corresponding to the best quality of life and 30 to the worst. Negative numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with either psoriasis or psoriatic arthritis and evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoriasis | Psoriatic Arthritis
Number analyzed (Participants) | 55 | 49
units on a scale | -8.6 (9.0) | -5.5 (7.93)

7. Secondary Outcome: Mean Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Score at 12 Months in Participants With Ankylosing Spondylitis and Participants With Psoriatic Arthritis With Axial Symptoms
Description: The Ankylosing Spondylitis Quality of Life (ASQoL) questionnaire is a disease-specific instrument designed to measure health related quality of life (HRQOL) in participants with AS. Participants answer yes/no to 18 items assessing the current impact of AS on their quality of life status. The total score ranges from 0 to 18, with lower scores representing better AS-specific quality of life. Negative numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with either ankylosing spondylitis and or psoriatic arthritis with axial symptoms and evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Psoriatic Arthritis With Axial Symptoms: Participants with psoriatic arthritis with axial symptoms
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis With Axial Symptoms
Number analyzed (Participants) | 58 | 19
units on a scale | -6.7 (6.3) | -6.4 (4.8)

8. Secondary Outcome: Mean Change From Baseline in Treatment Satisfaction Questionnaire for Medicine (TSQM) Version 1.4 Score at 12 Months
Description: The 14-item Treatment Satisfaction Questionnaire for Medication (TSQM) Version 1.4 is an instrument to show that adherence is expected to be related with participants' satisfaction with therapy and that such satisfaction can be a function of not only the effect of the treatment, but also the services offered. TSQM responses are used to derive scores for scales measuring effectiveness, side effects, convenience, and global satisfaction (based on participant evaluation over the last 2 to 3 weeks, or since last medication use). Scores for each of the 4 scales range from 0 to 100 with higher scores indicating a better state or outcome (e.g., greater perceived effectiveness or satisfaction). Positive numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 48 | 49 | 49 | 44 | 39 | 43
units on a scale
  Effectiveness: number analyzed (Participants) | 46 | 49 | 49 | 39 | 36 | 41
  Effectiveness | 7.1 (37.8) | 7.5 (39.0) | 4.8 (37.3) | 6.0 (34.0) | 3.9 (39.1) | 15.2 (41.2)
  Side effects: number analyzed (Participants) | 32 | 40 | 18 | 24 | 27 | 36
  Side effects | 2.3 (23.5) | 9.4 (22.3) | -0.9 (12.4) | 5.9 (18.8) | 11.1 (18.6) | 11.1 (24.2)
  Convenience: number analyzed (Participants) | 48 | 48 | 48 | 43 | 39 | 43
  Convenience | 10.8 (18.2) | 10.4 (22.5) | 9.7 (19.5) | 8.9 (13.3) | 7.1 (14.8) | 14.5 (16.5)
  Global satisfaction: number analyzed (Participants) | 48 | 48 | 48 | 44 | 39 | 43
  Global satisfaction | 7.6 (19.1) | 7.0 (20.1) | 1.8 (22.2) | 9.9 (20.5) | 5.8 (17.9) | 11.3 (22.8)

9. Secondary Outcome: Mean Change From Baseline in Total Satisfaction With Information About Medicines Scale (SIMS) Score at 12 Months
Description: The Satisfaction with Information about Medicines Scale (SIMS) assesses whether an individual has received enough information about a range of topics relating to prescribed medication. Participants are asked to rate the amount of information they have received using the following response scale: "too much", "about right", "too little", "none received", "none needed". Total satisfaction rating is obtained by summing the scores for each item. If the participant is satisfied that he/she has received a particular aspect of medication information (with a rating of "about right" or "none needed"), this is given a score of 1. If the participant is dissatisfied with the amount of information received (with a rating of "too much", "too little", or "none received"), this is scored 0. Total scores range from 0 to 17 with high scores indicating a high degree of overall satisfaction with the amount of medication information received. Positive numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 55 | 45 | 49 | 49 | 46 | 45
units on a scale | -0.3 (5.3) | 2.3 (5.0) | 1.4 (4.7) | -0.1 (5.4) | 0.4 (3.5) | 0.9 (5.7)

10. Secondary Outcome: Mean Change From Baseline in Total Morisky Medication Adherence Scale, 4 Questions (MMAS-4) Score at 12 Months
Description: The Morisky Medication Adherence Scale-4 (MMAS-4 ) is a 4-item self-reported measure of medication-taking behavior. It measures intentional and non-intentional non-adherence. The MMAS-4 score is the sum of four questions and ranges from 0 to 4: The coding is 0, 1 (low adherence), 2, 3 (moderate adherence) and 4 (high adherence). Positive numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 57 | 49 | 50 | 51 | 50 | 44
units on a scale | 0.12 (0.38) | -0.02 (0.83) | 0.14 (0.54) | -0.02 (0.32) | 0.04 (0.35) | 0.32 (1.01)

11. Secondary Outcome: Mean Change From Baseline in in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP) Score at 12 Months
Description: The WPAI-SHP is a questionnaire used to assess the effect of the participant's health problems on their ability to work and perform regular activities. Presenteeism indicates the percentage of impairment while working due to health problems. Absenteeism indicates the percentage of work time missed due to health problems. Total activity impairment (TAI) indicates the percentage of general (non-work) activity impairment due to health problems. Total work productivity impairment (TWPI) indicates the percentage of overall work impairment due to health problems. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity. Negative numbers indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with evaluable data; participants who were employed with available data at baseline and 12 months are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 60 | 49 | 54 | 53 | 54 | 46
units on a scale
  Presenteeism: number analyzed (Participants) | 33 | 30 | 32 | 34 | 31 | 41
  Presenteeism | -30.6 (25.2) | -20.7 (30.7) | -19.7 (28.0) | -35.0 (26.5) | -33.2 (30.2) | -13.2 (33.4)
  Absenteeism: number analyzed (Participants) | 29 | 22 | 30 | 25 | 28 | 30
  Absenteeism | -5.6 (28.4) | -16.8 (31.8) | -4.6 (24.1) | -9.6 (23.5) | -8.2 (27.8) | -10.8 (44.7)
  Total activity impairment | -30.2 (27.0) | -14.7 (35.7) | -18.5 (24.1) | -34.5 (28.9) | -33.3 (30.7) | -24.6 (34.1)
  Total work productivity impairment: number analyzed (Participants) | 28 | 22 | 29 | 23 | 27 | 28
  Total work productivity impairment | -4.8 (19.9) | -3.7 (13.1) | -1.1 (16.0) | -0.9 (10.5) | -3.2 (10.4) | -4.0 (28.1)

12. Secondary Outcome: Mean Change From the 12 Months Prior to Treatment With Adalimumab to the 12 Months After Beginning Treatment With Adalimumab in Health Resource Utilization: Number of Hospital Inpatient Days and Number of Sick Leave Days
Description: The number of hospital inpatient days over the 3 months preceding the first adalimumab administration was documented and multiplied by 4 to obtain an estimate of 12-month data. The 12-month total post-treatment hospital inpatient days was obtained by adding the values obtained at months 3, 6, 9, and 12. The number of sick leave days (in employed participants) over the 3 months preceding the first adalimumab administration was documented and multiplied by 4 to obtain an estimate of 12-month data. The 12-month total post-treatment sick leave days was obtained by adding the values obtained at months 3, 6, 9, and 12. Negative numbers indicate improvement from the prior 12 months.
Time Frame: 12 months prior to treatment start (Month 0 [baseline]) and 12 months after treatment start (total 24 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 72 | 62 | 67 | 71 | 65 | 58
days
  Number of hospital inpatient days | -2.56 (11.93) | -5.00 (17.36) | -1.25 (6.00) | -3.75 (18.41) | -3.68 (15.32) | -2.91 (9.10)
  Number of sick leave days: number analyzed (Participants) | 40 | 43 | 40 | 44 | 37 | 41
  Number of sick leave days | -5.10 (15.37) | -0.91 (32.37) | -1.55 (7.14) | -1.16 (8.00) | -22.00 (82.81) | -6.68 (37.29)

13. Secondary Outcome: Mean Change From the 12 Months Prior to Treatment With Adalimumab to the 12 Months After Beginning Treatment With Adalimumab in Health Resource Utilization: Number of Hospitalizations and Number of Sick Leaves
Description: The number of hospitalizations over the 3 months preceding the first adalimumab administration was documented and multiplied by 4 to obtain an estimate of 12-month data. The 12-month total hospitalizations were obtained by adding the values obtained at months 3, 6, 9, and 12. The number of sick leaves (in employed participants) over the 3 months preceding the first adalimumab administration was documented and multiplied by 4 to obtain an estimate of 12-month data. The 12-month total sick leaves were obtained by adding the values obtained at months 3, 6, 9, and 12. Negative numbers indicate improvement from the prior 12 months.
Time Frame: 12 months prior to treatment start (Month 0 [baseline]) and 12 months after treatment start (total 24 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: occurrences
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 72 | 62 | 67 | 71 | 65 | 58
occurrences
  Number of hospitalizations | -0.28 (1.15) | -1.06 (2.97) | -0.18 (0.83) | -0.15 (0.98) | -0.35 (1.33) | -0.45 (1.34)
  Number of sick leaves: number analyzed (Participants) | 40 | 43 | 40 | 44 | 37 | 41
  Number of sick leaves | -0.58 (1.66) | -1.19 (4.30) | -0.20 (0.88) | 0.05 (0.68) | -1.81 (9.73) | -0.54 (2.05)

14. Secondary Outcome: Mean Change From the 12 Months Prior to Treatment With Adalimumab to the 12 Months After Beginning Treatment With Adalimumab in Health Resource Utilization: Number of Outpatient Visits
Description: The number of outpatient visits to general practitioners, immune-mediated inflammatory disease specialists, ophthalmologists, gastroenterologists, dermatologists, rheumatologists, physiatrists, physiotherapists, and nurses over the 3 months preceding the first adalimumab administration was documented and multiplied by 4 to obtain an estimate of 12-month data. The 12-month total outpatient visits were obtained by adding the values obtained at months 3, 6, 9, and 12. Negative numbers indicate improvement from the prior 12 months.
Time Frame: 12 months prior to treatment start (Month 0 [baseline]) and 12 months after treatment start (total 24 months)
Population: All participants in the Full Analysis Set with evaluable data. Data were not collected for visits to physiatrists and physiotherapists in the Psoriasis Arm/Group, and for visits to physiatrists in the Rheumatoid Arthritis Arm/Group.
Measure: Mean (Standard Deviation); unit: occurrences
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 72 | 58 | 62 | 73 | 61 | 53
occurrences
  General practitioner: number analyzed (Participants) | 69 | 52 | 46 | 68 | 58 | 49
  General practitioner | -4.32 (6.78) | -4.35 (6.32) | -2.97 (5.18) | -3.41 (4.47) | -5.06 (8.29) | -3.68 (5.56)
  Immune-mediated inflammatory disease specialist: number analyzed (Participants) | 64 | 41 | 46 | 53 | 55 | 41
  Immune-mediated inflammatory disease specialist | -2.02 (4.45) | -5.97 (6.99) | -2.93 (4.76) | -1.60 (4.41) | -2.76 (5.90) | -3.53 (4.83)
  Ophthalmologist: number analyzed (Participants) | 61 | 30 | 41 | 50 | 49 | 38
  Ophthalmologist | -0.35 (1.59) | 0.18 (1.59) | -0.44 (2.09) | 0.02 (0.15) | -0.15 (1.12) | -0.15 (1.32)
  Gastroenterologist: number analyzed (Participants) | 59 | 58 | 41 | 52 | 51 | 53
  Gastroenterologist | -0.40 (1.41) | -6.83 (7.33) | -0.33 (1.12) | -0.14 (0.91) | -0.13 (1.02) | -5.45 (8.27)
  Dermatologist: number analyzed (Participants) | 60 | 30 | 62 | 55 | 51 | 43
  Dermatologist | 0.13 (0.54) | -0.06 (1.95) | -5.71 (5.41) | -0.93 (2.08) | -0.02 (1.04) | -0.26 (2.26)
  Rheumatologist: number analyzed (Participants) | 72 | 31 | 43 | 73 | 61 | 39
  Rheumatologist | -6.18 (6.06) | -0.35 (2.37) | -1.16 (2.74) | -5.36 (4.90) | -7.96 (5.71) | 0.15 (1.98)
  Physiatrist: number analyzed (Participants) | 60 | 29 | 0 | 51 | 0 | 36
  Physiatrist | -0.04 (0.47) | 0.06 (0.24) |  | -0.09 (0.61) |  | 0.16 (0.85)
  Physiotherapist: number analyzed (Participants) | 59 | 28 | 0 | 52 | 49 | 35
  Physiotherapist | -0.33 (6.43) | 1.18 (4.85) |  | -0.75 (5.20) | -1.49 (9.62) | 0.00 (1.19)
  Nurse: number analyzed (Participants) | 64 | 49 | 41 | 55 | 50 | 47
  Nurse | -0.98 (3.30) | -1.75 (4.73) | -0.11 (0.68) | -0.96 (2.63) | -1.09 (3.64) | 0.00 (4.35)

15. Secondary Outcome: Mean Change From Baseline in Disease Activity Score 28 (DAS28) at 12 Months
Description: The Disease Activity Score 28 (DAS28) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity (on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. Negative values indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with either psoriatic arthritis with peripheral symptoms or rheumatoid arthritis and evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Psoriatic Arthritis With Peripheral Symptoms: Participants with psoriatic arthritis and peripheral symptoms
Arm/Group | Psoriatic Arthritis With Peripheral Symptoms | Rheumatoid Arthritis
Number analyzed (Participants) | 42 | 56
units on a scale | -3.4 (1.3) | -2.8 (1.6)

16. Secondary Outcome: Mean Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS ESR) at 12 Months
Description: The Ankylosing Spondylitis Disease Activity Score (ASDAS) tool is a self-administered questionnaire/objective laboratory evaluation. The questionnaire assesses disease activity, back pain, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and duration of morning stiffness on a numeric rating scale (from 0 to 10, with 0 being none and 10 representing a duration of ≥2 hours). The laboratory parameter is a measurement of erythrocyte sedimentation rate (mm/hour; ESR). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and ESR) are combined to yield a score (0 to no defined upper limit). Negative values indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with either ankylosing spondylitis or psoriatic arthritis with axial symptoms and evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis With Axial Symptoms
Number analyzed (Participants) | 53 | 5
units on a scale | -1.6 (1.7) | -2.0 (1.4)

17. Secondary Outcome: Mean Change From Baseline in Clinical Disease Activity Index (CDAI) Score at 12 Months
Description: The Crohn's Disease Activity Index (CDAI) is a research tool used to quantify the symptoms of patients with Crohn's disease. Participants were asked to record the frequency of stools, abdominal pain and general well-being on a daily basis. In addition to the diary data, the investigator assessed the following for the calculation of CDAI: presence of complications (arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. The CDAI is the sum of the products of each item multiplied by a weighting factor and generally ranges from 0 up to 600, where remission of Crohn's disease is defined as CDAI < 150, and severe disease is defined as CDAI > 450. Negative values indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with Crohn's disease and evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 48
units on a scale | -174.9 (95.3)

18. Secondary Outcome: Mean Change From Baseline in Partial Mayo (pMayo) Score at 12 Months
Description: The Partial Mayo score (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). Negative values indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with ulcerative colitis and evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ulcerative Colitis
Number analyzed (Participants) | 45
units on a scale | -4.8 (2.6)

19. Secondary Outcome: Mean Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at 12 Months
Description: The Psoriasis Area and Severity Index (PASI) is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Negative values indicate improvement from baseline.
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with psoriasis and evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoriasis
Number analyzed (Participants) | 56
units on a scale | -16.6 (8.6)

20. Secondary Outcome: Participants' Rating of the AbbVie Care 2.0 Program at 12 Months
Description: All participants enrolled in the study were enrolled in the AbbVie Care 2.0 patient support (PSP) program. Participants rated the PSP program as either "Very good", "good", "less satisfying" or "I do not use the services" at the last study visit.
Time Frame: 12 months
Population: All participants in the Full Analysis Set with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 62 | 50 | 54 | 56 | 50 | 45
Participants
  Very good | 39 | 20 | 28 | 33 | 31 | 28
  Good | 20 | 28 | 23 | 22 | 19 | 16
  Less Satisfying | 3 | 2 | 1 | 1 | 0 | 0
  I do not use the services | 0 | 0 | 2 | 0 | 0 | 1

21. Secondary Outcome: Correlation Between Disease Activity Scores and Disease-specific Quality of Life Scores
Description: To define possible correlations between disease activity scores and disease specific quality of life scores, correlation analyses were performed. Correlation between patient socio-demographics, patient type and indication was not completed because these were uninterpretable per protocol.
  ASQoL= Ankylosing Spondylitis Quality of Life questionnaire
  ASDAS(ESR) = Ankylosing Spondylitis Disease Activity Score; laboratory parameter is a measurement of erythrocyte sedimentation rate (mm/hour; ESR)
  DAS28(ESR)= Disease Activity Score 28; laboratory parameter is a measurement of erythrocyte sedimentation rate (mm/hour; ESR)
  SIBDQ= Short Quality of Life in Inflammatory Bowel Disease Questionnaire
  CDAI= Clinical Disease Activity Index
  DLQI= Dermatology Life Quality Index
  PASI= Psoriasis Area and Severity Index
  pMayo= Partial Mayo score (Mayo score without endoscopy)
Time Frame: Baseline (Month 0) and 12 months
Population: All participants in the Full Analysis Set with evaluable data
Measure: Number; unit: correlation coefficient
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 54 | 45 | 55 | 13 | 46
correlation coefficient
  ASQoL - ASDAS(ESR): number analyzed (Participants) | 54 | 0 | 0 | 0 | 0
  ASQoL - ASDAS(ESR) | -0.213 |  |  |  |
  ASQoL - DAS28(ESR): number analyzed (Participants) | 0 | 0 | 0 | 13 | 0
  ASQoL - DAS28(ESR) |  |  |  | 0.132 |
  SIBDQ - CDAI: number analyzed (Participants) | 0 | 45 | 0 | 0 | 0
  SIBDQ - CDAI |  | -0.138 |  |  |
  DLQI - PASI: number analyzed (Participants) | 0 | 0 | 55 | 0 | 0
  DLQI - PASI |  |  | 0.323 |  |
  SIBDQ - pMayo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 46
  SIBDQ - pMayo |  |  |  |  | -0.453

22. Secondary Outcome: Correlation Between the Length of AbbVie Care 2.0 Duration and Participant Outcomes
Description: The effectiveness of the AbbVie Care 2.0 patient care support program (PSP) on participant outcomes was to be analyzed by applying mixed linear models on outcomes including PSP utilization (continuous vs terminated) as fixed variables. Baseline participant outcome values were also to be included in the model.
Time Frame: From Baseline (Month 0) to 12 months
Population: Assessment of the effectiveness of the length of PSP exposure on participant outcomes was not possible because of the low number of participants in the non-PSP group.
Arm/Group | Ankylosing Spondylitis | Crohn's Disease | Psoriasis | Psoriatic Arthritis | Rheumatoid Arthritis | Ulcerative Colitis
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent serious adverse events (TESAEs) were collected from the time of study drug administration until 70 days after the last dose of study drug (up to 62 weeks).
Description: TESAEs were collected whether elicited or spontaneously reported by the participant. Nonserious adverse events were not collected in this study.
Arm/Group | Adalimumab and AbbVie Care 2.0
All-Cause Mortality (participants affected / at risk) | 2/412
Serious Adverse Events (participants affected / at risk) | 19/412
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab and AbbVie Care 2.0 (N=412)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 3 (3)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (1)
DEATH (General disorders) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1)
HOSPITALIZATION (Surgical and medical procedures) | 1 (1)
TONSILLECTOMY (Surgical and medical procedures) | 1 (1)
SYNCOPE (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The key limitation of the study is the absence of a control group (participants treated with adalimumab without AbbVie Care 2.0). Given this limitation it is difficult to measure the impact of adding AbbVie Care 2.0 to adalimumab on study outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT02750800/Prot_SAP_000.pdf